CLINICAL TRIAL: NCT04543760
Title: Effect of Prone Positioning Combined With High Flow Oxygen Therapy on Oxygenation During Acute Respiratory Failure Due to Sars-covid-2: a Randomized Crossover Trial.
Brief Title: Effect of Prone Positioning Combined With High Flow Oxygen Therapy on Oxygenation During Acute Respiratory Failure Due to COVID-19
Acronym: DeCOPO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital St. Joseph, Marseille, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2020-04-03
Record Dates: First submitted 2020-09-08; First posted 2020-09-10 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Prone Position; Supine Position

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- [PP sequence 1] - Wash-out - [SP sequence 2] (Other)
  Interventions: Other: Prone position; Other: Supine position
- [SP sequence 1] - Wash-out - [PP sequence 2] (Other)
  Interventions: Other: Prone position; Other: Supine position

INTERVENTIONS:
Other: Prone position — prone positioning in spontaneous ventilation
Other: Supine position — supine positiong in spontaneous ventilation

SUMMARY:
The main manifestation of COVID-19 is acute hypoxemic respiratory failure (AHRF). In patients with AHRF, the need for invasive mechanical ventilation is associated with high mortality.

Prone positioning (PP) is a recommended strategy for patients with moderate to severe acute respiratory distress syndrome (ARDS) undergoing invasive mechanical ventilation.

Early PP combined with High Flow Oxygen Therapy may benefit spontaneous breathing patients with AHRF due to COVID-19 as recently reported in Jiangsu.

Our hypothesis is that early PP combined with High Flow Oxygen Therapy in patients with AHRF due to COVID-19 improves oxygenation.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years,
* Admitted to ICU within 72 hours,
* Having confirmed or highly suspected COVID-19 infection (positive RT-PCR and/or computed tomography),
* Having acute hypoxemic respiratory failure with a [PaO2/FiO2] ratio between 100 mmHg and 300 mmHg,
* Having given free and informed written consent,
* Being affiliated with or benefiting from a social security scheme.

Exclusion Criteria:

* Unable to achieve a prone position for mobility reasons,
* Unable to achieve a prone position due to agitation whatever the cause,
* With clinical occlusive syndrome in order to limit the risk of inhalation,
* Having a contraindication to the use of the esophageal catheter,
* Having signs of respiratory distress or disturbance of consciousness requiring intubation within the next hours,
* Having hypercapnia indicating the use of non-invasive ventilation (PaO2> 50 mmHg),
* Having severe hypoxemia defined by PaO2 / FiO2 <100mmHg,
* Ongoing pregnancy or breastfeeding,
* Subject to a measure for the protection of justice.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-01-15 (Actual); Study Completion 2021-03-14 (Actual)

PRIMARY OUTCOMES:
[PaO2 / FiO2] ratio | 6 hours
  Oxygenation will be evaluated by the [PaO2 / FiO2] ratio, measured at the beginning (baseline) and at the end of each 2h-sequence by arterial gasometry. The values of this ratio in PP and SP will be compared with each other.

SECONDARY OUTCOMES:
ΔPeso measured using an esophageal balloon catheter | 6 hours
  ΔPeso (cm H2O): defined at each inspiratory cycle as the difference between the esophageal pressure at the end of expiration and at the end of inspiration.
Concentration of CO2 at the end of expiration (EtCO2, mmHg) | 6 hours
  Capnometry measurements by breathing on a mouthpiece connected to an online analyzer.
  The measurements will be made on a 2 min recording (analysis of the curves over a period of 1 min) at the end of each sequence (PP or SP) and compared with each other.
Intensity of dyspnea | 6 hours
  assessed by the visual analogue scale for dyspnea (collected at the beginning and at the end of each 2h sequence; the values at the end of each sequence will be compared with each other): 0 = no breathlessness to 10 = worst breathlessness possible
Tolerance of the technique | 6 hours
  measured by the visual analogue scale for pain (collected at the beginning and at the end of each 2h-sequence; the values at the end of each sequence will be compared with each other): 0 = no pain to 10 = worst pain possible
Tolerance of the technique | 6 hours
  measured by the visual analogue scale for discomfort (collected at the beginning and at the end of each 2h-sequence; the values at the end of each sequence will be compared with each other): 0 = no discomfort to 10 = worst discomfort possible
The occurrence of side effects due to PP | 6 hours
  Oxygen desaturation (SaO2 <90%), occurrence of hemodynamic instability (Systolic blood pressure <80 mmHg or heart rate >120 mmHg for >1 minute), accidental withdrawal of venous catheter central or peripheral, accidental withdrawal of arterial catheter, accidental withdrawal of urinary catheter.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel LEHINGUE, M.D, Principal Investigator — Hopital Saint Joseph Marseille
Locations (4):
- France (4):
  - Hopital Européen, Marseille
  - Hopital La Timone, Marseille
  - Hopital Saint Joseph, Marseille
  - Hopital Nord, Marseille

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the published article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol
Time Frame: beginning 3 months and ending 2 years following article publication
Access Criteria: The data will be shared with investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose.
  The proposal should be directed to the PI, Dr Lehingue.